CLINICAL TRIAL: NCT06180577
Title: A Retrospective Survey Study to Assess the Accessibility, Preference, and Frequency of Adolescents Using Nerivio in School Setting
Brief Title: A Survey Study to Assess the Accessibility of the Nerivio Device At School
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE007
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-02

CONDITIONS: Migraine in Children
Keywords: Migraine; Nerivio; Headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adolescent Nerivio Users: Adolescent with migraine who used Nerivio at least once
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — Nerivio is a prescribed Remote Electrical Neuromodulation (REN) device for treatment of migraine

SUMMARY:
This is a retrospective survey-study to assess the accessibility, preference, and frequency of adolescents using Nerivio by itself, in combination with pharmacological medications, or not at all, in the school setting. The study population is prescribed Nerivio users, under the age of 18 years old, who have used the Nerivio device at least once. The study will be conducted electronically, and will include eligibility questions, an electronic informed consent form signed by the parent/legal guardian (e-ICF), an assent form signed by the adolescent patient (e-Assent), and an e-survey relating to the management of headaches due to migraine attacks. Participants will be recruited from Nerivio's userbase and will be compensated for their participation.

DETAILED DESCRIPTION:
This is a retrospective survey-study to assess the accessibility, preference, and frequency of adolescents using Nerivio by itself, in combination with pharmacological medications, or not at all, in the school setting. The study population is prescribed Nerivio users, under the age of 18 years old, who have used the Nerivio device at least once.

Study group: Participants will be recruited from Nerivio's user database. An invitation message will be sent via emails and/or in-app notifications to Nerivio users who are (1) under the age of 18 years old, and (2) treated with Nerivio at least once. Adolescents who meet these criteria will be invited to answer a screening questionnaire verifying eligibility.

Adolescents who are found eligible will be offered the opportunity to participate in the study. If they are willing, they will first be directed to an Informed Consent Form (e-ICF) to be signed by the participant's parent/legal guardian. A copy of the completed form will be automatically sent to the parent/legal guardian upon completion. If the parent/legal guardian consents via the e-ICF to his/her child's participation, an electronic assent form will follow and must be signed by the adolescent patient. A copy of the assent form will be automatically sent to the parents and the adolescent patient. Once both electronic consent forms are signed, the adolescent patient will be enrolled in the study and will be directed to the study survey.

Primary outcome measures:

Percent of adolescents' who prefer treating headaches due to migraine when they are at school with Nerivio alone, relative to other options (combination, pharmaceutical, not treating while in school).

Secondary outcome measures:

1. - Distribution of barriers to adolescents who report the necessity to treat their headaches due to migraine while at school, including the need to leave class for treatment, lack of availability of treatments while at school, and time delay to treat headaches.
2. - Distribution of treatments used by adolescents at school to treat migraine headaches prior to being prescribed Nerivio (specific pharmaceutical agents, or not treating at all) reflecting convergence to using Nerivio at school.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤18 years old at registration to the Nerivio app
* Treated with Nerivio at least once (≥30 minutes/treatment).
* Attended elementary, middle, junior high, or high school, while first prescribed Nerivio
* Must obtain parent/legal guardian consent form prior to signing the assent form by the adolescent and engaging in study survey.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with migraine who used Nerivio at least once
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Nerivio usage at school | 1 year
  Percent of adolescents who prefer treating headaches due to migraine when they are at school with Nerivio alone, relative to other options (combination, pharmaceutical, not treating while in school).

SECONDARY OUTCOMES:
Limitations to migraine treatment at school | 1 year
  Distribution of barriers to adolescents who report the necessity to treat their headaches due to migraine while at school, including need to leave class for treatment, lack of availability of treatments while at school, time delay to treat headaches.
Types of migraine treatments during school | 1 year
  Distribution of treatments used by adolescents at school to treat migraine headaches prior to being prescribed Nerivio (specific pharmaceutical agents, or not treating at all) reflecting convergence to using Nerivio at school.

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark Inbar, PhD, Study Director — Theranica Bio-Electronics Ltd
Locations (1):
- Theranica USA Inc, Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No